CLINICAL TRIAL: NCT00227773
Title: Phase II Study of Vatalanib and Octreotide in Patients With Progressive Low-Grade Neuroendocrine Tumors
Brief Title: Vatalanib and Octreotide in Treating Patients With Progressive Neuroendocrine Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000446076; ECOG-E6203
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Gastrointestinal Carcinoid Tumor; Islet Cell Carcinoma
Keywords: localized gastrointestinal carcinoid tumor; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; regional gastrointestinal carcinoid tumor; recurrent islet cell carcinoma; gastrinoma; insulinoma; WDHA syndrome; glucagonoma; pancreatic polypeptide tumor; somatostatinoma
MeSH Terms: conditions — Carcinoma, Islet Cell; Gastrinoma; Insulinoma; Vipoma; Glucagonoma; Somatostatinoma | interventions — Octreotide; vatalanib; Biological Therapy

INTERVENTIONS:
Drug: octreotide acetate
Drug: vatalanib
Procedure: anti-cytokine therapy
Procedure: antiangiogenesis therapy
Procedure: biological therapy
Procedure: endocrine therapy
Procedure: enzyme inhibitor therapy
Procedure: growth factor antagonist therapy
Procedure: hormone therapy
Procedure: protein tyrosine kinase inhibitor therapy
Procedure: somatostatin analogue therapy

SUMMARY:
RATIONALE: Vatalanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by stopping blood flow to the tumor. Octreotide may help control symptoms, such as diarrhea, caused by the tumor. Giving vatalanib together with octreotide may be an effective treatment for neuroendocrine tumors.

PURPOSE: This phase II trial is studying how well giving vatalanib together with octreotide works in treating patients with progressive neuroendocrine tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 4-month progression-free and overall survival of patients with progressive low-grade neuroendocrine tumors treated with vatalanib and octreotide.
* Determine the response rate in patients treated with this regimen.
* Determine the effect of this regimen on tumor markers (e.g., chromogranin A, 5-HIAA, and gastrin) in these patients.
* Determine the toxicity and tolerability of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral vatalanib once daily on days 1- 28 and octreotide* intramuscularly or IV on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients on a stable dose (i.e., no changes in dosage within the past 3 months) of octreotide before study entry remain on their current dose and schedule during study participation; patients who experience hypersensitivity and/or toxicity to octreotide may receive vatalanib alone.

After completion of study treatment, patients are followed at 4 weeks, every 3 months for 2 years, and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 23-44 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed low-grade neuroendocrine tumors
* The following tumor types are excluded:
* Small cell lung cancer
* Medullary thyroid cancer
* Paraganglioma
* Pheochromocytoma
* Measurable disease
* Radiographic evidence of disease progression after completion of any prior systemic therapy, chemoembolization, bland embolization, or observation within the past year, defined as either of the following:
* Appearance of a new lesion
* At least 20% increase in the longest diameter (LD) of any previously documented lesion or an increase in the sum of the LDs of multiple lesions in the aggregate of 20%

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 8.0 g/dL

Hepatic

* Bilirubin ≤ 2.0 times upper limit of normal (ULN)
* AST ≤ 3 times ULN (5 times ULN if liver metastases are present)

Renal

* Creatinine ≤ 1.5 times ULN
* Meets 1 of the following criteria:
* Urine protein negative by dipstick
* Urine protein:creatinine ratio < 1.0
* Urine protein < 1 g by 24-hour urine collection

Gastrointestinal

* Must be able to swallow tablets
* No ulcerative disease
* No uncontrolled nausea, vomiting, or diarrhea
* No bowel obstruction
* No other gastrointestinal tract disease resulting in an inability to take oral medication

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must be able to receive a contrast-enhanced CT scan
* No known history of allergic reaction to vatalanib or its derivatives or octreotide injections

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 4 weeks since prior chemotherapy
* No more than 1 prior systemic chemotherapy regimen
* Chemoembolization is not considered systemic chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 3 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* At least 4 weeks since prior major surgery

Other

* At least 4 weeks since other prior systemic therapy
* At least 4 weeks since prior local liver therapy
* No prior anti-vascular endothelial growth factor agents
* No concurrent grapefruit or grapefruit juice
* No concurrent therapeutic warfarin or similar oral anticoagulants that are metabolized by the cytochrome P450 system
* Concurrent heparin allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Holen, MD, Study Chair — University of Wisconsin, Madison; Mary Mulcahy, MD — Robert H. Lurie Cancer Center